CLINICAL TRIAL: NCT03290183
Title: Confocal Laser Endomicroscopy in Pleural Malignancies: A Comparison With Pathology
Brief Title: Confocal Laser Endomicroscopy in Pleural Malignancies
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Prof J.T. Annema, Head of pulmonary endoscopy department, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: NL60800.018.17
Record Dates: First submitted 2017-08-24; First posted 2017-09-21 (Actual); Last update posted 2017-09-21 (Actual); Status verified 2017-09

CONDITIONS: Pleural Malignant Mesothelioma; Thymoma; Pleural Diseases
Keywords: Confocal laser endomicroscopy
MeSH Terms: conditions — Mesothelioma, Malignant; Thymoma; Pleural Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intrathoracic malignancy: Patients with (strong suspicion of) intrathoracic malignancy and an indication for tissue collection by CT-guided, transthoracic or thoracoscopic approach undergo additional imaging with confocal laser endomicroscopy (CLE).
  Interventions: Device: Confocal laser endomicroscopy

INTERVENTIONS:
Device: Confocal laser endomicroscopy — Real-time microscopic imaging technique
  Other Names: CLE

SUMMARY:
To date, the different biopsy methods, such as CT-guided pleural biopsy, mediastinal biopsy, endosonography and thoracoscopy have their limitations in diagnosing pleural malignancies, such as mesothelioma. Sampling errors frequently occur resulting in the common histological finding of 'non-specific pleuritic/fibrosis', which presents a great uncertainty for clinicians and patients. Confocal laser endomicroscopy (CLE) provides real-time imaging on a cellular level, however data of CLE in pleural malignancies are lacking.

DETAILED DESCRIPTION:
Novel optical imaging techniques such as confocal laser endomicroscopy (CLE) have emerged in recent years as techniques that actually enable in vivo real-time microscopic analysis of malignancies of the GI-tract and lung cancer. Through recent advances the probe became small enough to fit through a biopsy needle and can be used during CT-guided and endosonographic guided biopsies (EUS-FNA). Patients with intra-thoracic malignancies often require invasive procedures such as bronchoscopy, thoracoscopy, mediastinoscopy, transthoracic needle aspiration or surgical exploration to obtain a diagnosis. Intra thoracic malignancies encompass lung cancers, thymomas and malignant pleural mesothelioma. These tumors often present with pleural thickening, unilateral pleural effusion, mediastinal enlargement or a peripheral located mass in the lungs. Tissue collection of the suspected pleural thickening is required to assess a diagnosis and differentiate between the tumor types, to classify and to stage in a proper manner. To date, the different biopsy methods, such as CT-guided pleural biopsy, mediastinal biopsy, endosonography and thoracoscopy have their limitations in diagnosing these malignancies. Sampling errors frequently occur resulting in the common histological finding of 'non-specific pleuritic/fibrosis', which presents a great uncertainty for clinicians and patients. Novel microscopic imaging techniques such as CLE are capable of real time imaging on a cellular level. Data of CLE in intra-thoracic malignancies are lacking.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Supected intra-thoracic malignancies with pleural involvement and referred for a diagnostic procedure by thoracoscopy, CT guided biopsy or endosonography

Exclusion Criteria:

* Inability and willingness to provide informed consent
* Patients with known allergy for fluorescein or risk factors for an allergic reaction
* pregnancy or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspected intra-thoracic malignancies, who are referred for diagnostic work-up by either transthoracic, thoracoscopic or endosonographic biopsy.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2017-08-28 (Actual); Primary Completion 2018-08-28 (Estimated); Study Completion 2019-03-01 (Estimated)

PRIMARY OUTCOMES:
Technical feasibility: Number of successful procedures with evaluable CLE-imaging | cross sectional (1 day)
  Number of successful procedures with evaluable CLE-imaging
Procedure-related adverse events | cross sectional (1 day)
  Number of study-related adverse events
To describe and develop visual descriptive image criteria (number of descriptive criteria based on CLE imaging) | cross sectional (1 day)
  Qualitative description of the number of descriptive criteria based on CLE imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Jouke Annema, MD,PhD, Principal Investigator — Department of respiratory medicine, Academic Medical Center Amsterdam
Locations (2):
- Netherlands (2):
  - Academic Medical Center, Amsterdam, Noordd-Holland
  - NKI-AvL, Amsterdam, North Holland

IPD SHARING:
Plan to Share IPD: Yes
CLE imaging